CLINICAL TRIAL: NCT05705856
Title: Effectiveness and Safety of Ustekinumab Intensification in Crohn's Disease: a Retrospective Observational Study
Brief Title: Effectiveness and Safety of Ustekinumab Intensification in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0004
Record Dates: First submitted 2023-01-15; First posted 2023-01-31 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease
Keywords: ustekinumab; dose escalation; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- intravenous maintenance at early stage: Participants who have evidence of high activity clinically, biochemically or endoscopically : HBI ≥8, inflammatory markers significantly increased (CRP > 5mg/L, fecal calprotectin> 200mg/g), SES-CD≥ 7, will get multiple intravenous injections of Ustekinumab maintenance after induction.
  Interventions: Drug: Ustekinumab
- intravenous escalation when poor response: Participants who experience a loss of response or poor response to 90 mg Ustekinumab standard therapy will receive Ustekinumab intravenously at regular interval or at shorten interval.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Patients will receive an intravenous induction (adjusted 6 mg/kg dose) followed by subcutaneous 90 mg every 12 or 8 weeks, and will receive dose escalation when response is not effective enough.
  Other Names: UST; Ustekinumab antibody

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of intravenous administration at regular intervals of Ustekinumab in participants with loss of response to standard regimen or have evidence of high activity clinically, biochemically or endoscopically.

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of intravenous administration at regular intervals of Ustekinumab. It consists of escalation treatment period (Week 0 to 52); and safety follow up visit (24 weeks after last dose). Study assessments will include Harvey-Bradshaw index (HBI), Physician Global Assessment Score (PGA), laboratory evaluations, endoscopic evaluation, review of concomitant medications and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* With active Crohn's disease
* Undergoing Ustekinumab dose intensification with at least two or more intravenous infusions at the discretion of the treating physician
* HBI ≥ 5 before Ustekinumab therapy
* Over 18 years of age

Exclusion Criteria:

* Who had received Ustekinumab for an indication
* Pregnant or nursing
* L4 type
* History of enterectomy or enterostomy related to disease
* Who used total enteral nutrition for more than 2 weeks due to complications such as obstruction, abscess and perforation after starting Ustekinumab therapy
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Ustekinumab dose intensification with at least two or more intravenous infusions at the discretion of the treating physician instead of a scheduled SC dose at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with steroid-free clinical remission at Week 24 | Week24
  Percentage of participants with steroid-free clinical remission at Week 24 from the escalation will be assessed. Steroid-free clinical remission (performed only in patients on prednisone or budesonide at time of initiation of UST) was defined as tapering off steroids completely and HBI ≤ 4 points or complete resolution in CD symptoms or severity assessed by PGA.

SECONDARY OUTCOMES:
Percentage of participants with biochemical remission at Week 24 | Week 24
  Percentage of participants with biochemical remission at Week 24 from the escalation will be assessed. Biochemical remission was defined as a CRP concentration ≤5 mg/L and a FCP level of ≤200 µg/g.
Percentage of participants with endoscopic remission at Week 52 | Week 52
  Percentage of participants with endoscopic remission at Week 52. Endoscopic remission was defined as SES-CD ≤3 or absence of ulcers or described as the absence of ulceration.
Percentage of participants with normal fecal calprotectin level at Week 52 | Week 52
  Percentage of participants with normal fecal calprotectin level at 52w (among patients with baseline fecal calprotectin greater than 200ug/g)
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 1.5 years
  The percentage of participants with at least one adverse event and subcategories of adverse events will be assessed. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Percentage of Participants with Infections and Serious Infections | up to 1.5 years
  Percentage of participants with infections and serious infections will be reported.
Percentage of Participants continue UST | up to 1.5 years
  Proportion of patients who continue UST during the follow-up will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No